CLINICAL TRIAL: NCT01681615
Title: Challenge Test for Acetylsalicylic Acid Hypersensitivity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: University Hospital, Akershus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: ASA-ST-OS; 2012-000698-22 (EudraCT Number)
Record Dates: First submitted 2012-08-09; First posted 2012-09-10 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Asthma Aspirin-sensitive; ASA Intolerant Asthma; Asthma, Aspirin-Induced; Asthma, Nasal Polyps, and Aspirin Intolerance
Keywords: Challenge test for Aspirin Hypersensitivity; Challenge test for Acetylsalicylic Hypersensitivity
MeSH Terms: conditions — Asthma, Aspirin-Induced; Asthma, Nasal Polyps, And Aspirin Intolerance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetylsalicylate (Active Comparator): Acetylsalicylic Acid Eyedrops
  Interventions: Drug: Acetylsalicylate
- isotonic NaCl (Placebo Comparator): Saline Eyedrops
  Interventions: Drug: Isotonic NaCl

INTERVENTIONS:
Drug: Acetylsalicylate — 1-2 drops
  Arms: Acetylsalicylate
Drug: Isotonic NaCl — 1 drop
  Arms: isotonic NaCl

SUMMARY:
The investigators want to find new challenge test for Acetylsalicylic hypersensitivity / Aspirin hypersensitivity. The investigators suggest that this new test will be as efficient as the already established protocols in terms of sensitivity and specificity.

DETAILED DESCRIPTION:
Hypersensitivity to Acetylsalicylic Acid or Aspirin (and other NSAIDS) is a condition that affects up to 2,5% of the population. Most cases are seen in a complex of such hypersensitivity with chronic eosinophilic rhinosinusitis with nasal polyposis and asthma. Despite research in finding a reliable in-vitro-test for the condition, challenge tests are still considered gold standard. So far oral, nasal, inhalation and intravenous routes of administration has been described in literature.

ELIGIBILITY:
Inclusion Criteria:

* Persons between 18 and 60 years of age
* Suspected Acetylsalicylic Acid Hypersensitivity

Exclusion Criteria:

* History on anaphylactic shock after NSAIDS intake
* History on gastric ulcer after NSAIDS intake
* Patients previously gone through testing or desensitisation for Aspirin hypersensitivity
* Clinical unstable asthma or baseline FEV1<70%
* Severe disease of the heart, digestive tract, liver or kidney
* Severe chronic urticaria
* Present conjunctivitis
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-03 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Inspiratory nasal flow measured by Rhinomanometry | Within 45 min from challenge
  Bilateral flow reduction >40% considered positive test.
Expiratory nasal flow measured by Rhinomanometry | Within 45 min from challenge
  Bilateral expiratory flow reduction >40% considered positive.
Pulmonary forced expiratory volume in 1 second (FEV1) | Within 45 min from challenge
  Reduction in FEV1 >20% is considered as positive test.

SECONDARY OUTCOMES:
Conjunctival symptoms | Within 45 days from challenge
  0=no symptoms, 1=limited redness and / or itching, 2=conjunctival redness and /or itching / swelling or bullae within 5 minutes from testing.
  Value 1 and 2 is considered positive if unilateral.
Nasal symptoms | Within 45 minutes from challenge
  Rhinorrhea, congestion and sneezing is considered as positive test.
Bronchial and laryngeal symptoms | Within 45 minutes from challenge
  Bronchospasm. tight chest, wheezing or laryngospasm is considered as positive test.

OTHER OUTCOMES:
Other significant and relevant symptoms | Within 45 days after challenge
  Erythema in upper body or face, nausea or abdominal pain is considered as positive test.

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Bachmann-Harildstad, MD, PhD, Study Chair — University in Oslo
Locations (2):
- Norway (2):
  - Akershus University Hospital, Lørenskog, Akershus
  - Stavanger University Hospital, Stavanger, Rogaland

REFERENCES:
- [Background] Stevenson DD, Sanchez-Borges M, Szczeklik A. Classification of allergic and pseudoallergic reactions to drugs that inhibit cyclooxygenase enzymes. Ann Allergy Asthma Immunol. 2001 Sep;87(3):177-80. doi: 10.1016/S1081-1206(10)62221-1. No abstract available. PMID 11570612
- [Background] Hedman J, Kaprio J, Poussa T, Nieminen MM. Prevalence of asthma, aspirin intolerance, nasal polyposis and chronic obstructive pulmonary disease in a population-based study. Int J Epidemiol. 1999 Aug;28(4):717-22. doi: 10.1093/ije/28.4.717. PMID 10480701
- [Background] Kasper L, Sladek K, Duplaga M, Bochenek G, Liebhart J, Gladysz U, Malolepszy J, Szczeklik A. Prevalence of asthma with aspirin hypersensitivity in the adult population of Poland. Allergy. 2003 Oct;58(10):1064-6. doi: 10.1034/j.1398-9995.2003.00267.x. PMID 14510727
- [Background] Vally H, Taylor ML, Thompson PJ. The prevalence of aspirin intolerant asthma (AIA) in Australian asthmatic patients. Thorax. 2002 Jul;57(7):569-74. doi: 10.1136/thorax.57.7.569. PMID 12096197
- [Background] Samter M, Beers RF Jr. Intolerance to aspirin. Clinical studies and consideration of its pathogenesis. Ann Intern Med. 1968 May;68(5):975-83. doi: 10.7326/0003-4819-68-5-975. No abstract available. PMID 5646829
- [Background] Stevenson D SR, Zuraw BL. Sensitivity to aspirin and NSAIDs. Adkinson NJ YJ, Busse WW, et al., editor. Philadelphia: CV Mosby and Co.; 2003
- [Background] Nizankowska-Mogilnicka E, Bochenek G, Mastalerz L, Swierczynska M, Picado C, Scadding G, Kowalski ML, Setkowicz M, Ring J, Brockow K, Bachert C, Wohrl S, Dahlen B, Szczeklik A. EAACI/GA2LEN guideline: aspirin provocation tests for diagnosis of aspirin hypersensitivity. Allergy. 2007 Oct;62(10):1111-8. doi: 10.1111/j.1398-9995.2007.01409.x. Epub 2007 May 22. PMID 17521312
- [Background] Mastalerz L, Setkowicz M, Sanak M, Szczeklik A. Hypersensitivity to aspirin: common eicosanoid alterations in urticaria and asthma. J Allergy Clin Immunol. 2004 Apr;113(4):771-5. doi: 10.1016/j.jaci.2003.12.323. PMID 15100686
- [Background] Setkowicz M, Mastalerz L, Podolec-Rubis M, Sanak M, Szczeklik A. Clinical course and urinary eicosanoids in patients with aspirin-induced urticaria followed up for 4 years. J Allergy Clin Immunol. 2009 Jan;123(1):174-8. doi: 10.1016/j.jaci.2008.09.005. Epub 2008 Oct 8. PMID 18842291
- [Background] Szczeklik A, Gryglewski RJ, Czerniawska-Mysik G. Relationship of inhibition of prostaglandin biosynthesis by analgesics to asthma attacks in aspirin-sensitive patients. Br Med J. 1975 Jan 11;1(5949):67-9. doi: 10.1136/bmj.1.5949.67. PMID 1109660
- [Background] Wong JT, Nagy CS, Krinzman SJ, Maclean JA, Bloch KJ. Rapid oral challenge-desensitization for patients with aspirin-related urticaria-angioedema. J Allergy Clin Immunol. 2000 May;105(5):997-1001. doi: 10.1067/mai.2000.104571. PMID 10808182
- [Background] Berges-Gimeno MP, Simon RA, Stevenson DD. Long-term treatment with aspirin desensitization in asthmatic patients with aspirin-exacerbated respiratory disease. J Allergy Clin Immunol. 2003 Jan;111(1):180-6. doi: 10.1067/mai.2003.7. PMID 12532116
- [Background] Rozsasi A, Polzehl D, Deutschle T, Smith E, Wiesmiller K, Riechelmann H, Keck T. Long-term treatment with aspirin desensitization: a prospective clinical trial comparing 100 and 300 mg aspirin daily. Allergy. 2008 Sep;63(9):1228-34. doi: 10.1111/j.1398-9995.2008.01658.x. PMID 18699939
- [Background] Stevenson DD. Aspirin sensitivity and desensitization for asthma and sinusitis. Curr Allergy Asthma Rep. 2009 Mar;9(2):155-63. doi: 10.1007/s11882-009-0023-4. PMID 19210906
- [Background] Stevenson DD, Hankammer MA, Mathison DA, Christiansen SC, Simon RA. Aspirin desensitization treatment of aspirin-sensitive patients with rhinosinusitis-asthma: long-term outcomes. J Allergy Clin Immunol. 1996 Oct;98(4):751-8. doi: 10.1016/s0091-6749(96)70123-9. PMID 8876550
- [Background] Sweet JM, Stevenson DD, Simon RA, Mathison DA. Long-term effects of aspirin desensitization--treatment for aspirin-sensitive rhinosinusitis-asthma. J Allergy Clin Immunol. 1990 Jan;85(1 Pt 1):59-65. doi: 10.1016/0091-6749(90)90222-p. PMID 2299107
- [Background] Macy E, Bernstein JA, Castells MC, Gawchik SM, Lee TH, Settipane RA, Simon RA, Wald J, Woessner KM; Aspirin Desensitization Joint Task Force. Aspirin challenge and desensitization for aspirin-exacerbated respiratory disease: a practice paper. Ann Allergy Asthma Immunol. 2007 Feb;98(2):172-4. doi: 10.1016/S1081-1206(10)60692-8. PMID 17304886
- [Background] Romano A, Torres MJ, Castells M, Sanz ML, Blanca M. Diagnosis and management of drug hypersensitivity reactions. J Allergy Clin Immunol. 2011 Mar;127(3 Suppl):S67-73. doi: 10.1016/j.jaci.2010.11.047. PMID 21354502
- [Background] Wismol P, Putivoranat P, Buranapraditkun S, Pinnobphun P, Ruxrungtham K, Klaewsongkram J. The values of nasal provocation test and basophil activation test in the different patterns of ASA/NSAID hypersensitivity. Allergol Immunopathol (Madr). 2012 May-Jun;40(3):156-63. doi: 10.1016/j.aller.2010.12.011. Epub 2011 Apr 13. PMID 21492991
- [Background] Alonso-Llamazares A, Martinez-Cocera C, Dominguez-Ortega J, Robledo-Echarren T, Cimarra-Alvarez M, Mesa del Castillo M. Nasal provocation test (NPT) with aspirin: a sensitive and safe method to diagnose aspirin-induced asthma (AIA). Allergy. 2002 Jul;57(7):632-5. doi: 10.1034/j.1398-9995.2002.t01-1-13447.x. PMID 12100305
- [Background] Milewski M, Mastalerz L, Nizankowska E, Szczeklik A. Nasal provocation test with lysine-aspirin for diagnosis of aspirin-sensitive asthma. J Allergy Clin Immunol. 1998 May;101(5):581-6. doi: 10.1016/S0091-6749(98)70163-0. PMID 9600492
- [Background] Krane Kvenshagen B, Jacobsen M, Halvorsen R. Can conjunctival provocation test facilitate the diagnosis of food allergy in children? Allergol Immunopathol (Madr). 2010 Nov-Dec;38(6):321-6. doi: 10.1016/j.aller.2010.01.007. Epub 2010 Jun 4. PMID 20605314
- [Background] Kralinger MT, Hamasaki D, Kieselbach GF, Voigt M, Parel JM. Intravitreal acetylsalicylic acid in silicone oil: pharmacokinetics and evaluation of its safety by ERG and histology. Graefes Arch Clin Exp Ophthalmol. 2001 Mar;239(3):208-16. doi: 10.1007/s004170100255. PMID 11405070
- [Background] Kralinger MT, Stolba U, Velikay M, Egger S, Binder S, Wedrich A, Haas A, Parel JM, Kieselbach GF. Safety and feasibility of a novel intravitreal tamponade using a silicone oil/acetyl-salicylic acid suspension for proliferative vitreoretinopathy: first results of the Austrian Clinical Multicenter Study. Graefes Arch Clin Exp Ophthalmol. 2010 Aug;248(8):1193-8. doi: 10.1007/s00417-010-1389-7. Epub 2010 Apr 28. PMID 20424852
- [Background] Voigt M, Kralinger M, Kieselbach G, Chapon P, Anagnoste S, Hayden B, Parel JM. Ocular aspirin distribution: a comparison of intravenous, topical, and coulomb-controlled iontophoresis administration. Invest Ophthalmol Vis Sci. 2002 Oct;43(10):3299-306. PMID 12356838